CLINICAL TRIAL: NCT07150949
Title: A Prospective Randomized Phase II Trial of Long-Course Chemoradiotherapy or Short-Course Radiotherapy Combined With CAPOX, PD-1 Antibody, and a COX-2 Inhibitor for Microsatellite Stable Locally Advanced Rectal Cancer (SERRAC)
Brief Title: Long-course Chemoradiotherapy or Short-course Radiotherapy Combined With CAPOX, PD-1antibody, and COX-2 Inhibitor for MSS Locally Advanced Rectal Cancer (SERRAC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-2025-254-4403
Record Dates: First submitted 2025-08-27; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Locally Advanced Rectal Cancer; Neoadjuvant Therapy
MeSH Terms: interventions — Oxaliplatin; Capecitabine; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-course Radiotherapy plus chemotherapy group (Experimental)
  Interventions: Radiation: Long-course radiotherapy; Drug: Oxaliplatin; Drug: Capecitabine; Drug: Celecoxib; Drug: Serplulimab
- Short-course Radiotherapy plus immunochemotherapy group (Experimental)
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Celecoxib; Radiation: Short-course radiotherapy; Drug: Serplulimab

INTERVENTIONS:
Radiation: Long-course radiotherapy — Long-course radiation: 50Gy/25Fx
  Other Names: LCRT
  Arms: Long-course Radiotherapy plus chemotherapy group
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w
Drug: Capecitabine — Xeloda
Drug: Celecoxib — celecoxib 200 mg orally twice a day
Radiation: Short-course radiotherapy — Short-course radiotherapy: 25Gy/5Fx
  Other Names: SCRT
  Arms: Short-course Radiotherapy plus immunochemotherapy group
Drug: Serplulimab — Serplulimab 300mg, d1, q3w

SUMMARY:
SERRAC is a prospective, multicentre, randomized phase II trial. 138 LARC (T3-4/N+M0, distance from anal verge ≤10cm) patients will be treated with neoadjuvant therapy and assigned to Group A and Group B (1:1). Group 1 receives LCRT (50Gy/25Fx) followed by 3 cycles of CAPOX.Group 2 receives SCRT (25Gy/5Fx) followed by 4 cycles of capecitabine plus oxaliplatin (CAPOX) chemotherapy and PD-1 antibody. The COX2 inhibitor celecoxib 200 mg was started orally twice a day during chemotherapy until the end of neoadjuvant treatment.TME surgery is scheduled after TNT while a watch and wait (W&W) option can be applied to patients achieving clinical complete response (cCR). The primary endpoint is complete response (CR, pathological complete response [pCR] plus cCR) rate. The secondary endpoints include the grade 3-4 acute adverse effects (AE) rate, anal preservation rate, 3-year DFS rate, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years, gender not limited
2. Pathologically confirmed rectal adenocarcinoma
3. ≤10 cm from the anus
4. Baseline stage T3-4/N+
5. No distant metastasis
6. MSI/MMR status MSS/pMMR
7. Karnofsky performance status score ≥70
8. No prior chemotherapy or other anti-cancer treatment prior to enrollment
9. No prior immunotherapy prior to enrollment
10. Ability to comply with the study protocol
11. Written informed consent

Exclusion Criteria:

1. Pregnancy or breast-feeding women;
2. Known history of other malignancies within 5 years;
3. Known history of previous anti-tumor treatment, including radiotherapy, chemotherapy, immune checkpoint inhibitors, T cell-related therapy, etc;
4. Known history of severe neurological or mental illness (such as schizophrenia, dementia or epilepsy);
5. Current severe cardiac disease (cardiac dysfunction and arrhythmia), renal dysfunction and liver dysfunction;
6. Acute cardiac infarction or cerebral ischemic stroke occurred within 6 months before recruitment;
7. Uncontrolled infection which needs systemic therapy;
8. Active autoimmune disease or immunodeficiencies, known history of organ transplantation or systematic use of immunosuppressive agents;
9. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV 1 to 2 antibody positive), active syphilis infection, active pulmonary tuberculosis infection
10. Allergic to any component of the therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate | 1 month after the surgery or the decision of W&W
  Rate of complete response (CR), including the rate of pathologic complete response (pCR) after surgery and the rate of cCR with W&W strategy.

SECONDARY OUTCOMES:
Grade 3-4 adverse effects rate | From date of randomization until 3 months after the completion neoadjuvant therapy
  Rate of chemotherapy, radiotherapy and immunotherapy related adverse events
3 year anal preservation rate | From date of randomization until the date of or date of death from any cause, whichever came first, assessed up to 36 months.
  3 year anal preservation rate
3 year disease free survival rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months.
  Rate of 3 year disease free survival
3 year local recurrence free survival rate | From date of randomization until the date of first documented pelvic failure, assessed up to 36 months.
  Rate of 3 year local recurrence free survival
3 year overall survival rate | From date of randomization until the date of death from any cause, assessed up to 36 months.
  Rate of 3 year overall survival
Rate of surgical complications | The surgical complications were assessed within 3 months after the surgery.
  Rate of surgical complications, such as intraoperative hemorrhage, anastomotic leakage, intestinal obstruction, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, M.D, PH.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China